CLINICAL TRIAL: NCT00783224
Title: Comparative Study of Mometasone Furoate Nasal Spray and Fluticasone Propionate Nasal Spray in Patients With Perennial Allergic Rhinitis
Brief Title: A Comparative Study of Mometasone Furoate Nasal Spray and Fluticasone Propionate Nasal Spray in Patients With Perennial Allergic Rhinitis (Study P04512)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P04512
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2010-07-12 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate; Fluticasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mometasone Furoate Placebo (PLAMF) (Placebo Comparator): Placebo to mometasone furoate nasal spray, made to be indistinguishable from mometasone furoate nasal spray
  Interventions: Drug: Placebo for MF
- Fluticasone Propionate Placebo (PLAFP) (Placebo Comparator): Placebo to fluticasone propionate nasal spray, made to be indistinguishable from fluticasone propionate nasal spray
  Interventions: Drug: Placebo for FP
- Mometasone Furoate (MF) (Experimental): Mometasone furoate nasal spray 200 μg/day(QD)
  Interventions: Drug: Mometasone
- Fluticasone Propionate (FP) (Active Comparator): Fluticasone Propionate nasal spray 200 μg/day, twice per day (BID)
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Placebo for MF — Placebo to mometasone furoate nasal spray, indistinguishable from mometasone furoate nasal spray. Patients in this arm take 2 sprays per nostril once a day for 2 weeks
  Arms: Mometasone Furoate Placebo (PLAMF)
Drug: Placebo for FP — Placebo to fluticasone nasal spray, indistinguishable from fluticasone propionate nasal spray. Patients in this arm take 2 sprays per nostril twice a day for 2 weeks
  Arms: Fluticasone Propionate Placebo (PLAFP)
Drug: Mometasone — Mometasone furoate nasal spray. Patients in this arm take 2 sprays per nostril once a day for 2 weeks
  Other Names: SCH 032088; Nasonex
  Arms: Mometasone Furoate (MF)
Drug: Fluticasone — Fluticasone propionate nasal spray. Patients in this arm take 2 sprays per nostril twice a day for 2 weeks
  Other Names: Flonase
  Arms: Fluticasone Propionate (FP)

SUMMARY:
This study was conducted to see if mometasone nasal spray is efficaceous for the treatment of perennial allergic rhinitis. Patients will be randomized to active mometasone, placebo mometasone, active fluticasone, or placebo fluticasone.

ELIGIBILITY:
Inclusion Criteria:

Patients with perennial allergic rhinitis meeting all of the followings.

* Patients with symptoms of perennial allergic rhinitis, the severity of which is moderate or severer according to the severity grading provided in the "Guidelines for the Management of Allergic Rhinitis in Japan" (partly modified) with the 4-nasal symptom score of 4 or over at informed consent and during the pre-treatment observation period
* Patients with positive reaction to the eosinophil count in nasal discharge or nasal challenge test in addition to the skin test or specific IgE antibody test
* Outpatients aged 16 years or over at informed consent
* Patients in either sex
* Patients (or their legal representatives in case of patients aged under 20 years) capable of giving written informed consent
* Patients capable of recording nasal allergy diary every day

Exclusion Criteria:

* Patients with a complication of tuberculous diseases or lower respiratory tract infections, and those with a complication of otorhinolaryngeal infections(acute upper respiratory tract inflammation, acute laryngopharyngitis, acute tonsillitis, etc.) requiring treatments judged by the investigator (subinvestigator) at the time of enrollment to randomization
* Patients with a complication of infection or systemic mycosis for which no effective antibiotics are available
* Patients with a complication of recurrent epistaxis
* Patients with uncured nasal septal ulcer, operated nose or nasal trauma.
* Patients with a history of hypersensitivity to steroids and any ingredients of the study drugs
* Pregnant, lactating or possibly pregnant patients or the patients who themselves or whose partners wish to become pregnant during the study
* Patients with severe hepatic or renal disorder, heart or blood disease, diabetes mellitus, hypertension, or other serious complication, suffering from problems with systemic condition
* Patients who have pollens as multiple allergens and the period from 7 days before enrollment to randomization to completion of the treatment period coincides with the period of scattering of relevant pollens
* Patients with a complication of vasomotor rhinitis or eosinophilic rhinitis
* Patients with a complication of a nasal disease (infectious sinusitis, hypertrophic rhinitis, acute or chronic rhinitis, nasal polyps, or septal deviation) which may interfere with efficacy evaluation of the study drugs
* Patients with a complication of a disease (acute upper respiratory tract inflammation, acute laryngitis or acute tonsillitis, etc.) of severity affecting nasal symptoms within 7 days before enrollment
* Patients who have previously received MF nasal spray
* Patients who used FP nasal spray within 28 days before initiation of the pre-treatment observation period (7 days before enrollment to randomization)
* Patients who have participated in clinical trials of other investigational product(s) within 120 days (4 months) before obtaining informed consent or participating at present
* Patients in whom prior medication expected to be effective for allergic rhinitis was not drawn long enough before initiation of treatment with the investigational product or the preceding medication cannot be withdrawn
* Patients who are being treated with specific desensitization therapy or nonspecific allassotherapy or in whom such the therapy was withdrawn within 90 days (3 months) before obtaining informed consent (except for patients receiving the maintenance therapy at present in whom the therapy began more than 180 days (6 months) before obtaining the informed consent)
* Other patients whom the investigator or the subinvestigator judged to be inappropriate for participation in the present study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-12 (Actual)

REFERENCES:
- [Result] N. Sou et. al; Allergology & Immunology 16(3) page 394-413, (2009.02) -Japanese language journal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mometasone Furoate Placebo (PLAMF) | Fluticasone Propionate Placebo (PLAFP) | Mometasone Furoate (MF) | Fluticasone Propionate (FP)
Started | 32 | 34 | 143 | 142
Completed | 32 | 34 | 142 | 140
Not Completed | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Discarded the Investigational Drug Used | 0 | 0 | 0 | 1
Not completed — Inappropriate as a study subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Placebo (PLAMF) | Fluticasone Propionate Placebo (PLAFP) | Mometasone Furoate (MF) | Fluticasone Propionate (FP) | Total
Number analyzed (Participants) | 32 | 34 | 143 | 142 | 351
Age, Customized [Number; unit: participants]
  <20 years old | 1 | 0 | 7 | 11 | 19
  20-29 years old | 20 | 13 | 59 | 76 | 168
  30-39 years old | 11 | 16 | 54 | 33 | 114
  40-59 years old | 0 | 5 | 19 | 21 | 45
  >=60 years old | 0 | 0 | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 99 | 87 | 230
  Male | 12 | 10 | 44 | 55 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change in 4 Nasal Symptom Score (Sneezing Attack, Rhinorrhea, Nasal Congestion, and Nasal Itching) After 2 Weeks
Description: The nasal symptoms (sneezing attacks, rhinorrhea, nasal congestion and itching) were rated in 4 grades (+++: 3 points, ++: 2 points, +: 1 point, -: 0 point) based on the evaluation criteria for nasal symptoms. Total possible best score is 0 points, total possible worst score is 12 points.
Time Frame: Baseline to 2 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mometasone Furoate Placebo (PLAMF) | Fluticasone Propionate Placebo (PLAFP) | Mometasone Furoate (MF) | Fluticasone Propionate (FP)
Number analyzed (Participants) | 32 | 34 | 143 | 142
Units on a scale
  Baseline | 7.84 (0.25) | 8.41 (0.29) | 8.27 (0.15) | 8.29 (0.16)
  Two Weeks | 1.63 (0.37) | 1.74 (0.35) | 3.90 (0.17) | 3.69 (0.17)
Statistical Analysis 1: Comparison: Mometasone Furoate Placebo (PLAMF) vs Mometasone Furoate (MF); Test type: Superiority or Other; p = 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Placebo (PLAFP) vs Fluticasone Propionate (FP); Test type: Superiority or Other; p = 0.0001, ANCOVA

ADVERSE EVENTS:
Groups:
- Mometasone Furoate Placebo and Fluticasone Propionate Placebo: Both placebo groups (arms) were combined to report adverse events
Arm/Group | Mometasone Furoate Placebo and Fluticasone Propionate Placebo | Mometasone Furoate (MF) | Fluticasone Propionate (FP)
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/143 | 1/142
Other Adverse Events (participants affected / at risk) | 4/66 | 11/143 | 4/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Placebo and Fluticasone Propionate Placebo (N=66) | Mometasone Furoate (MF) (N=143) | Fluticasone Propionate (FP) (N=142)
Wisdom Teeth Removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Placebo and Fluticasone Propionate Placebo (N=66) | Mometasone Furoate (MF) (N=143) | Fluticasone Propionate (FP) (N=142)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only restriction on the PI is that the PI needs to get approval from the sponsor for publication of the trial results prior to public release.